CLINICAL TRIAL: NCT02125929
Title: Comparative Study of the Efficacy and Safety Outcomes of Robotic, Laparoscopic and Open Surgery for Enucleation of Benign Pancreatic Neuroendocrine Tumors
Brief Title: Comparative Study of Robotic, Laparoscopic and Open Surgery for Enucleation of Benign Pancreatic Neoplasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHGS2013; ENRLO (Other: Peking Union Medical College Hospital)
Record Dates: First submitted 2014-04-26; First posted 2014-04-29 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Pancreatic Neuroendocrine Tumors
MeSH Terms: interventions — Robotic Surgical Procedures; Laparoscopy; Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- robotic arm (Experimental): robotic surgery for enucleation benign Pancreatic Neuroendocrine Tumors Case number = 50
  Interventions: Procedure: Robotic surgery
- Laparoscopic surgery (Experimental): laparoscopic surgery for enucleation benign Pancreatic Neuroendocrine Tumors Case number = 50
  Interventions: Procedure: Laparoscopic surgery
- Open surgery (Experimental): Open surgery for enucleation benign Pancreatic Neuroendocrine Tumors Case number = 100
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: Robotic surgery — Robotic surgery: enucleation benign Pancreatic Neuroendocrine Tumors
  Arms: robotic arm
Procedure: Laparoscopic surgery — Laparoscopic surgery: enucleation benign Pancreatic Neuroendocrine Tumors
  Arms: Laparoscopic surgery
Procedure: Open surgery — Open surgery: enucleation benign Pancreatic Neuroendocrine Tumors
  Arms: Open surgery

SUMMARY:
To determine the efficacy and safety of robotic, laparoscopic and open surgery for enucleation of benign pancreatic neuroendocrine tumors

DETAILED DESCRIPTION:
The study was prospective and retrospective, non-randomized study included patients with benign pancreatic neoplasms. The robotic arm consecutively includes patients underwent robotic enucleation surgery and expected number in this arm is 50. The laparoscopic and open surgery arms retrospectively include case from the year 2004. The number of patients for laparoscopic and open surgery arms are 50 and 100, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Body Mass Index<30
* Preoperative diagnosis of resectable benign Pancreatic Neuroendocrine Tumors
* Tumor type: Non-functional pancreatic endocrine tumours and insulinomas
* largest diameter < 4cm
* Preoperative CT showed no evidence that tumor was connected with main pancreatic duct

Exclusion Criteria:

* Severe cardio/pulmonary complications
* Other pancreatic diseases, including pancreatitis and pancreatic cancer
* Multiple pancreatic neuroendocrine tumors
* Distant metastasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pancreatic fistula rate | up to 30 days

SECONDARY OUTCOMES:
Mortality rate | up to 30 days

OTHER OUTCOMES:
Intra-operative bleeding volume | intra operative
Operation Time | Intra operative
Conversion rate to open surgery | Intra operative
  Only applied to the robotic surgery arm and laparoscopic arm
Quality of life and pain scores | up to 30 days
Delayed gastric emptying rate | up to 30 days
Intra-abdominal bleeding rate | up to 30 days
Postoperative infection rate | up to 30 days
Hospital stay time | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yupei Zhao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of General Surgery, Peking Union medical school hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tian F, Hong XF, Wu WM, Han XL, Wang MY, Cong L, Dai MH, Liao Q, Zhang TP, Zhao YP. Propensity score-matched analysis of robotic versus open surgical enucleation for small pancreatic neuroendocrine tumours. Br J Surg. 2016 Sep;103(10):1358-64. doi: 10.1002/bjs.10220. Epub 2016 Aug 2. PMID 27480993